CLINICAL TRIAL: NCT00501891
Title: A Phase II Study of Bevacizumab in Combination With Metronomic Temozolomide for Recurrent Malignant Glioma
Brief Title: Bevacizumab in Combination With Metronomic Temozolomide for Recurrent Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000404; AVF3821s; P04860
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-03

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme; Brain and Central Nervous System Tumors; Recurrent Malignant Glioma; Recurrent Glioblastoma Multiforme; Avastin; Bevacizumab; Temodar; Temozolomide
MeSH Terms: conditions — Glioblastoma; Central Nervous System Neoplasms; Glioma | interventions — Bevacizumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab and Metronomic Temozolomide (Experimental): Patients will receive up to 12 cycles of bevacizumab (Avastin) and metronomic temozolomide (Temodar), and each cycle is 28 days. Bevacizumab will be administered at 10 mg/kg every other week beginning a minimum of 7 days after a biopsy or 28 days after a craniotomy. Temozolomide will be dosed at 50 mg/m2 daily in a 28-day cycle.
  Interventions: Drug: Bevacizumab; Drug: Metronomic Temozolomide

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab administered intravenously 10mg/kg every other week.
  Other Names: Avastin
Drug: Metronomic Temozolomide — Temozolomide 50mg/m2 given orally on a daily basis.
  Other Names: Temodar

SUMMARY:
This is a phase II study of the combination of Avastin and metronomic temozolomide in recurrent malignant glioma patients. The primary objective will be to determine the efficacy of Avastin (bevacizumab) and metronomic temozolomide in malignant glioma patients. The secondary objective will be to determine the safety of Avastin, 10 mg/kg every other week, in combination with metronomic temozolomide in terms of progression-free survival.

DETAILED DESCRIPTION:
This is a phase II trial of the combination of Avastin and metronomic temozolomide in recurrent WHO grade IV malignant glioma patients. Patients will receive up to 12 cycles of Avastin and temozolomide and cycles are continuous 28 days. Patients will receive daily temozolomide at a dose of 50mg/m2 and will receive Avastin every other week at a dose of 10mg/kg. Patients will be required to have a baseline MRI within 2 weeks of starting treatment and a repeat MRI every 8 weeks. A total of 32 patients will be enrolled at Duke.

Patients with recurrent malignant gliomas have a very poor prognosis, so new therapies are needed. Given the activity of metronomic temozolomide and the safety and activity of Avastin against malignant glioma, it is reasonable to study the combination in recurrent malignant glioma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of WHO grade IV primary malignant glioma
* Karnofsy Performance Status (KPS) >/= 60%
* Evidence of measurable primary CNS neoplasm on contrast-enhanced MRI.
* An interval of at least 4 weeks between prior surgical resection or 1 week from a biopsy and enrollment on this protocol
* An interval of at least 4 weeks from the end of prior radiotherapy or one week from the end of a cycle of chemotherapy and enrollment on this protocol.
* No evidence of CNS hemorrhage on the baseline MRI or CT scans

Exclusion Criteria:

* Life expectancy < 8 weeks
* Pregnancy or breast feeding
* Progression to metronomic temozolomide, defined as tumor progression while taking daily temozolomide or progression within 4 weeks of stopping metronomic temozolomide
* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center (Brain Tumor Center), Durham, North Carolina, United States

REFERENCES:
- [Result] Desjardins A, Reardon DA, Coan A, Marcello J, Herndon JE 2nd, Bailey L, Peters KB, Friedman HS, Vredenburgh JJ. Bevacizumab and daily temozolomide for recurrent glioblastoma. Cancer. 2012 Mar 1;118(5):1302-12. doi: 10.1002/cncr.26381. Epub 2011 Jul 26. PMID 21792866
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — http://cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab and Temozolomide: Patients will receive up to 12 cycles of Avastin and temozolomide, and each cycle is 28 days. Avastin will be administered at 10 mg/kg every other week beginning a minimum of 7 days after a biopsy or 28 days after a craniotomy. Temozolomide will be dosed at 50 mg/m2 daily in a 28-day cycle.
Period: Overall Study
Arm/Group | Bevacizumab and Temozolomide
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab and Temozolomide
Number analyzed (Participants) | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 54.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: 6-Month Progression-free Survival
Description: Percentage of participants surviving six months from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression according to the Macdonald criteria, or to death due to any cause. [Optional: Macdonald criteria are standard criteria in neuro-oncology. Tumor assessment was made according to the adapted MacDonald criteria based on the combined evaluation of: 1) assessment of the MRI scan for measurable, evaluable, and new lesions (made by the independent external expert too), 2) overall assessment of neurological performance (made by the investigator), 3) concomitant steroid use (as reported by the investigator).]
Time Frame: 6 months
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Bevacizumab and Metronomic Temozolomide: Patients will receive up to 12 cycles of Avastin and temozolomide, and each cycle is 28 days. Avastin will be administered at 10 mg/kg every other week beginning a minimum of 7 days after a biopsy or 28 days after a craniotomy. Temozolomide will be dosed at 50 mg/m2 daily in a 28-day cycle.
Arm/Group | Bevacizumab and Metronomic Temozolomide
Number analyzed (Participants) | 32
percentage of participants | 18.8 [7.6 to 33.7]

2. Secondary Outcome: Response Rate
Description: The number of participants with complete or partial response as determined by a modification of the Macdonald criteria. Complete response was defined as complete disappearance on MR/CT of all enhancing tumor and mass effect, off all corticosteroids (or receiving only adrenal replacement doses), accompanied by a stable or improving neurologic examination, and maintained for at least 4 weeks. Partial Response was defined as greater than or equal to 50% reduction in tumor size on MR/CT by bi-dimensional measurement, on a stable or decreasing dose of corticosteroids, accompanied by a stable or improving neurologic examination, and maintained for at least 4 weeks.
Time Frame: 27 months
Population: Intent to treat
Measure: Number; unit: Number of participants
Arm/Group | Bevacizumab and Metronomic Temozolomide
Number analyzed (Participants) | 32
Number of participants | 9

3. Secondary Outcome: Incidence and Severity of CNS Hemorrhage and Systemic Hemorrhage
Description: Number of participants experiencing a Central Nervous System (CNS) hemorrhage or systemic hemorrhage
Time Frame: 27 months
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Bevacizumab and Metronomic Temozolomide
Number analyzed (Participants) | 32
participants
  CNS Hemorrhage | 0
  Systemic Hemorrhage | 0

4. Secondary Outcome: Incidence of Grade ≥ 4 Hematologic or Grade ≥ 3 Non-hematologic Toxicity
Description: Number of participants experiencing a grade ≥4 hematologic or grade ≥3 non-hematologic toxicity
Time Frame: 27 months
Population: Intent to treat
Measure: Number; unit: participants
Groups:
- Bevacizumab and Metromonic Temozolomide: Patients will receive up to 12 cycles of Avastin and temozolomide, and each cycle is 28 days. Avastin will be administered at 10 mg/kg every other week beginning a minimum of 7 days after a biopsy or 28 days after a craniotomy. Temozolomide will be dosed at 50 mg/m2 daily in a 28-day cycle.
Arm/Group | Bevacizumab and Metromonic Temozolomide
Number analyzed (Participants) | 32
participants
  Grade ≥ 4 hematologic toxicities | 0
  Grade ≥ 3 non-hematologic toxicities | 14

ADVERSE EVENTS:
Time Frame: 27 months
Description: The adverse events were gather in Common Terminology Criteria for Adverse Events (CTCAE) v.3.0, and have been converted to v.4.0 for entry into ClinicalTrials.gov.
Arm/Group | Bevacizumab and Temozolomide
Serious Adverse Events (participants affected / at risk) | 8/32
Other Adverse Events (participants affected / at risk) | 15/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab and Temozolomide (N=32)
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 3
Lung infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab and Temozolomide (N=32)
Blurred vision (Eye disorders) | 6
Nausea (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 6
Ataxia (Nervous system disorders) | 5
Cognitive disturbance (Nervous system disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 4
Dysphasia (Nervous system disorders) | 3
Memory impairment (Nervous system disorders) | 6
Peripheral motor neuropathy (Nervous system disorders) | 6
Confusion (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 2
Sexual dysfunction, NOS (Reproductive system and breast disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No